CLINICAL TRIAL: NCT03713502
Title: The Role of Environmental Enteropathy on HIV Associated Diabetes
Brief Title: Enteropathy and Diabetes in HIV Patients
Acronym: REEHAD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Institute for Medical Research, Tanzania (Other Government)
Collaborators: University of Copenhagen (Other); London School of Hygiene and Tropical Medicine (Other); Queen Mary University of London (Other)
Responsible Party: Principal Investigator, Dr George PrayGod, Principal Research Scientist, National Institute for Medical Research, Tanzania
Other Study IDs: TMA2017GSF-1965
Record Dates: First submitted 2018-10-17; First posted 2018-10-19 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Diabetes; Environmental Enteropathy; HIV
Keywords: Pre-diabetes; Diabetes; HIV; Enteropathy; Inflammation; Microbial translocation; Endotoxin translocation; Insulin resistance; Visceral obesity; Incretin hormones; GLP-1; GLP-2; GIP
MeSH Terms: conditions — Diabetes Mellitus; Glucose Intolerance; Intestinal Diseases; Inflammation; Insulin Resistance; Obesity, Abdominal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood, stool and urine samples collected for analysis of enteropathy biomarkers
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Emerging data suggest that HIV-infected people have disproportionately higher risk of diabetes than HIV-uninfected people. Multiple factors may contribute to elevated diabetes risk including increased prevalence of conventional non-communicable diseases (NCDs) risk factors, use of some antiretroviral drugs regimens, and inflammation and immune activation secondary to environmental- and HIV-enteropathy. To date, enteropathy has been little studied in relation to HIV and diabetes in Sub-Saharan Africa. Enteropathy leads to systemic inflammation which may in turn result in insulin resistance and may reduce secretion of incretins, the gut hormones which stimulate synthesis and secretion of insulin. Both mechanisms could potentially result in higher diabetes risk in HIV patients. This study investigates the hypothesis that among HIV-infected patients environmental enteropathy increase the risk of diabetes. The findings of this study will provide information which could be used as a basis for developing clinical trials to address different aspects of environmental enteropathy in order to reduce the burden of diabetes among HIV-infected populations

DETAILED DESCRIPTION:
This study will investigate if enteropathy is associated with higher risk of diabetes in HIV patients using a cross-sectional study design. To implement it cost-efficiently, investigators will nest it to an ongoing cohort study which investigates risk factors for diabetes and other chronic diseases among HIV patients in Tanzania (the CICADA study) (NCT03106480).

The CICADA study recruited 1947 participants during 2016/2017. These will be followed- up during 2017/2018 and 2018/2019 by which point it is expected that about 1550 participants will be retained in the cohort. Data collection for the current study will coincide with the final CICADA study follow-up. Data on demography, socio-economic status, conventional non-communicable disease risk factors, HIV and TB status, antiretroviral therapy use history, anthropometry, body composition, lipid profile, CD4 count, C-reactive protein, alpha-1-acid glycoprotein, insulin, and diabetes status will be retrieved from CICADA study. Data on gut enteropathy biomarkers i.e plasma citrulline, GLP-1, glucagon like peptide-2 (GLP-2), glucose-dependent insulinotropic polypeptide (GIP), fecal myeloperoxidase (MPO), neopterin, and alpha-1-antitrypsin, intestinal permeability (by 4-sugar test), lipopolysaccharide binding protein, tumor necrosis factor-α receptor, interleukin 6, and fecal elastase (as an indicator of pancreatic function) will be collected solely for this study to investigate the study hypothesis.

Data will be entered in Cspro and managed and analysed in STATA. Both linear and logistic regression will be used to assess the associations between exposure variables (markers of enteropathy) and outcome (diabetes). In addition, causal inference techniques will be used to investigate associations between enteropathy biomarkers and diabetes.

ELIGIBILITY:
Inclusion Criteria: Participants who were recruited in CICADA study (NCT03106480) during 2016/2017 and meet the following criteria:

* Aged 18 years or above
* HIV-infected
* HIV-uninfected
* Resident of Mwanza region
* Consent to take part in this study

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from HIV-infected patients attending antiretroviral therapy (ART) clinics in Mwanza (Tanzania) as well as from the general population (those who meet the inclusion criteria).
Sampling Method: Non-Probability Sample
Enrollment: 1947 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of diabetes | January 2019 to December 2019
  Investigators will determine prevalence of diabetes among participants with enteropathy and those without enteropathy
Prevalence of pre-diabetes | January 2019 to December 2019
  Investigators will determine prevalence of pre-diabetes among participants with enteropathy and those without enteropathy

CONTACTS AND LOCATIONS:
Overall Officials: Dr George PrayGod, MD, PhD, Principal Investigator — National Institute for Medical Research; Dr Daniel Faurholt-Jepsen, MD, PhD, Principal Investigator — University of Copenhagen; Prof Suzanne Filteau, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- NIMR Research Clinic, Mwanza, Mwanza Region, Tanzania

REFERENCES:
- [Background] Brown TT, Cole SR, Li X, Kingsley LA, Palella FJ, Riddler SA, Visscher BR, Margolick JB, Dobs AS. Antiretroviral therapy and the prevalence and incidence of diabetes mellitus in the multicenter AIDS cohort study. Arch Intern Med. 2005 May 23;165(10):1179-84. doi: 10.1001/archinte.165.10.1179. PMID 15911733
- [Background] Maganga E, Smart LR, Kalluvya S, Kataraihya JB, Saleh AM, Obeid L, Downs JA, Fitzgerald DW, Peck RN. Glucose Metabolism Disorders, HIV and Antiretroviral Therapy among Tanzanian Adults. PLoS One. 2015 Aug 19;10(8):e0134410. doi: 10.1371/journal.pone.0134410. eCollection 2015. PMID 26287742
- [Background] PrayGod G, Changalucha J, Kapiga S, Peck R, Todd J, Filteau S. Dysglycemia associations with adipose tissue among HIV-infected patients after 2 years of antiretroviral therapy in Mwanza: a follow-up cross-sectional study. BMC Infect Dis. 2017 Jan 30;17(1):103. doi: 10.1186/s12879-017-2209-z. PMID 28137307
- [Background] Prendergast A, Kelly P. Enteropathies in the developing world: neglected effects on global health. Am J Trop Med Hyg. 2012 May;86(5):756-63. doi: 10.4269/ajtmh.2012.11-0743. PMID 22556071
- [Background] Nazli A, Chan O, Dobson-Belaire WN, Ouellet M, Tremblay MJ, Gray-Owen SD, Arsenault AL, Kaushic C. Exposure to HIV-1 directly impairs mucosal epithelial barrier integrity allowing microbial translocation. PLoS Pathog. 2010 Apr 8;6(4):e1000852. doi: 10.1371/journal.ppat.1000852. PMID 20386714
- [Background] Klatt NR, Funderburg NT, Brenchley JM. Microbial translocation, immune activation, and HIV disease. Trends Microbiol. 2013 Jan;21(1):6-13. doi: 10.1016/j.tim.2012.09.001. Epub 2012 Oct 11. PMID 23062765
- [Background] Boden G. Free fatty acids, insulin resistance, and type 2 diabetes mellitus. Proc Assoc Am Physicians. 1999 May-Jun;111(3):241-8. doi: 10.1046/j.1525-1381.1999.99220.x. PMID 10354364
- [Background] James WP, Coore HG. Persistent impairment of insulin secretion and glucose tolerance after malnutrition. Am J Clin Nutr. 1970 Apr;23(4):386-9. doi: 10.1093/ajcn/23.4.386. No abstract available. PMID 5441174
- [Background] Indulekha K, Anjana RM, Surendar J, Mohan V. Association of visceral and subcutaneous fat with glucose intolerance, insulin resistance, adipocytokines and inflammatory markers in Asian Indians (CURES-113). Clin Biochem. 2011 Mar;44(4):281-7. doi: 10.1016/j.clinbiochem.2010.12.015. Epub 2011 Jan 8. PMID 21219897